CLINICAL TRIAL: NCT01053923
Title: A Feasibility Study of MRI in Assessment of Primary Tumor During Chemoradiation for Anal Canal and Perianal Cancer
Brief Title: MRI for Tumor During Chemoradiation for Anal Canal and Perianal Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Patient eligibility has limited accrual and patient sample has changed with the change in referral patients.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 09-0695-CE
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Anal Cancer Patients; Perianal Patients
Keywords: Perianal Cancer; Anal Cancer; MRI scan
MeSH Terms: conditions — Anus Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI Scan
  Interventions: Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — This study involves three imaging sessions (Magnetic Nuclear Resonance -MRI), with one session before radiation therapy and two sessions during radiation therapy (one at 3 weeks of RT; the other during the last week of RT). Each imaging session will last for approximately 45 to 60 minutes.

SUMMARY:
The purpose of this study is to establish a prospective database of anal canal and perianal cancer patients treated with IMRT and chemotherapy with curative intent at PMH for the purposes of investigating MRI-derived primary tumor parameters. Patients who decide to participate in this study will be treated according to standard treatment policies and radiation therapy planning protocols at Princess Margaret Hospital (PMH) with radiation therapy +/- chemotherapy. IMRT for all treatment phases of radiotherapy has been implemented as standard treatment. Surgery is reserved for salvage treatment.

DETAILED DESCRIPTION:
Anal cancer is an uncommon cancer, accounting for 2% of gastrointestinal cancers. Prognostic factors include tumor differentiation and staging, along with patient gender, race, and socioeconomic status. The standard of care is radical chemoradiation with 5-fluorouracil and mitomycin C, with surgery reserved for salvage. Intensity modulated radiation therapy (IMRT) is a specialized radiotherapy technique that may be used for anal cancer. IMRT allows the radiation dose to conform to the three-dimensional shape of the target volume more than conventional two-dimensional techniques, and it may reduce treatment toxicities without compromising tumor control. At the Princess Margaret Hospital (PMH) since July 2007, IMRT for all treatment phases of radiotherapy has been implemented as standard treatment for patients with anal canal and perianal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmation of invasive primary squamous cell carcinoma or adenocarcinoma of the anal canal or perianal region
* treatment with curative intent
* patients who are not eligible for chemotherapy and receive IMRT alone are eligible for evaluation
* primary anal or perianal cancer evaluable on cross-sectional imaging (CT or MRI) scan
* ECOG performance status of 0, 1, or 2
* age > 18 years
* able to provide informed consent

Exclusion Criteria:

* evidence of distant metastasis (M1)
* prior radiation therapy to the pelvis or contraindication to radiotherapy
* contraindication to MRI imaging
* known allergy to intravenous Gadolinium
* renal insufficiency (serum creatinine greater than 150)
* serious claustrophobia
* cardiac pacemaker
* hip prosthesis
* major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of imaging study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anal canal or perianal cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Primary tumor dimensions at simulation and during week 3 and last week of fractionated radiotherapy from MRI | 12 months
Primary tumor perfusion coefficient at simulation and during week 3 and last week of fractionated radiotherapy from MRI | 12 months
Primary tumor apparent diffusion coefficient at simulation and during week 3 and last week of fractionated radiotherapy from MRI | 12 months

SECONDARY OUTCOMES:
Change with time from start of radiotherapy course in primary tumor dimensions from MRI | 12 months
Change with time from start of radiotherapy course in primary tumor perfusion coefficient from MRI | 12 months
Change with time from start of radiotherapy course in primary tumor apparent diffusion coefficient from MRI | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dinniwell, MD, Principal Investigator — University Health Network, Princess Margaret Hospital